CLINICAL TRIAL: NCT04653987
Title: Ultrasound and Fluoroscopy Guided Percutaneous Transhepatic Biliary Drainage in Patients With Malignant Bile Duct Obstruction - Impact of Puncture Angle on Total Fluoroscopy Time Reduction
Brief Title: The Impact of Puncture Angle on Total Fluoroscopy Time Reduction During Percutaneous Biliary Drainage
Status: Completed | Type: Observational
Sponsor: Institut za Rehabilitaciju Sokobanjska Beograd (Other)
Collaborators: Klinički centar Srbije (Unknown)
Responsible Party: Principal Investigator, Tamara Filipovic, Phd, Institut za Rehabilitaciju Sokobanjska Beograd
Other Study IDs: 717/3
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Interventional Radiology
Keywords: biliary drainage, fluoroscopy time, puncture angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Puncture angle : ≤30 (group I) >30 (group II): The patients will be divided into two groups based on the puncture angle: ≤30° group and >30° group. The two groups will be retrospectively analyzed for technical success, fluoroscopy time and complications.
  Interventions: Procedure: Percutaneous biliary drainage
- Technical Parameters of all Interventions: Peripheral bile duct diameter, central bile duct diameter, number of punctures, type of drainage and total fluoroscopy time will be noted.
  Interventions: Procedure: Percutaneous biliary drainage

INTERVENTIONS:
Procedure: Percutaneous biliary drainage

SUMMARY:
The purpose of this study is to retrospectively assess the importance of initial bile duct puncture angle on total fluoroscopy time and overall efficacy during ultrasound and fluoroscopy guided percutaneous transhepatic biliary drainage (PTBD) performed for patients with malignant biliary hilar obstruction.

DETAILED DESCRIPTION:
Data used for this study will be collected from medical records of patients who underwent PTBD at the Interventional radiology department. Only patients who received percutaneous biliary drainage performed with right sided intercostal approach will be included in study. The initial puncture was ultrasound-guided in all patients. Any subsequent step of the procedure was performed under fluoroscopy. The cumulative fluoroscopy time (the total time of the exposure to X rays during intervention) after the US guided puncture was recorded. It will be used as an indirect measure of the complexity of the intervention and as an important parameter of radiation exposure. The patients will be divided into two groups based on the puncture angle: ≤30° group and >30° group. The two groups will be retrospectively analysed for technical success, fluoroscopy time and complications.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmation or imaging data confirming malignant disease causing bile duct obstruction, performance status 0-1.

Exclusion Criteria:

* terminally ill patiens, performance status ˃2, hepatic decompensation (including ascites), severe underlying cardiac or renal diseases and coagulation disorders

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with malignant biliary obstruction who underwent PTBD performed by right sided intercostal approach (US and fluorocopy guided).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Total fluoroscopy time | during intervention
  The initial puncture was ultrasound-guided in all patients. Any subsequent step of the procedure (PTBD) was performed under fluoroscopy. Total fluoroscopy time will be collected from Radiation Dose Report obtained in the angio suite workstation software ( General Electric Innova 540)

CONTACTS AND LOCATIONS:
Overall Officials: Dragan M Masulovic, Phd, Study Director — Clinical Centre of Serbia

IPD SHARING:
Plan to Share IPD: Undecided